CLINICAL TRIAL: NCT04610489
Title: Diagnostic Performance of an Antigen Test for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Infection (COVID-19)
Brief Title: Diagnostic Performance of an Antigen Test for SARS-CoV-2 Infection (COVID-19)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with recruiting for the study and with staffing the study.
Sponsor: Carilion Clinic (Other)
Responsible Party: Principal Investigator, John W Epling, Medical Director of Research, Department of Family Medicine, Carilion Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-20-1088; Epling-533 (Other: Carilion Clinic)
Record Dates: First submitted 2020-10-27; First posted 2020-10-30 (Actual); Results first posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Covid-19
Keywords: diagnostic test; antigen test; PCR test; symptomatic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Masking Description: simultaneous acquisition of both test of interest and reference standard without contingency
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Study Population (Other): All subjects will undergo bilateral mid-turbinate swabs for COVID Antigen (Quidel Sofia SARS Antigen Fluorescent Immunoassay (FIA)) as well as bilateral rt-PCR testing (Quest SARS-CoV-2 rRT-PCR).
  Interventions: Diagnostic Test: Quidel Sofia SARS Antigen FIA

INTERVENTIONS:
Diagnostic Test: Quidel Sofia SARS Antigen FIA — Obtained via bilateral mid-turbinate swab.

SUMMARY:
A comparison of a direct antigen test for SARS-CoV-2 obtained by mid-turbinate swab with the reference standard rt-PCR test obtained by nasopharyngeal swab in outpatients with symptoms compatible with COVID-19.

DETAILED DESCRIPTION:
This study plans to compare a direct antigen test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV2) obtained by mid-turbinate nasal swab with a reverse transcription polymerase chain reaction (rt-PCR) test obtained by nasopharyngeal swab (the current reference standard) in a population of patients with symptoms suggestive of COVID-19 for fewer than 5 days. Subjects whose physicians have already ordered an rt-PCR test at a Carilion testing center will be screened and recruited by phone during a required scheduling call. The study coordinator will describe the study by phone, and the subject will be consented when they arrive at the testing center. After consenting, a mid-turbinate swab direct antigen test will be obtained just prior to the ordered nasopharyngeal swab and any other ordered tests. The subjects will receive their rt-PCR test results through the usual channels of clinical notification. The subjects will not receive their nasal antigen results. The antigen test results will be analyzed in a batch process and the results entered into RedCap by the study staff. The rt-PCR results will be extracted from the Epic electronic health record using patient identifiers and paired with the corresponding antigen result for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Acutely ill with one or more COVID-19 symptoms

Exclusion Criteria:

* Unable to speak English
* Unable to provide written informed consent
* Symptoms have lasted longer than 5 days
* Currently hospitalized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John W Epling, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Clinic, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lambert-Niclot S, Cuffel A, Le Pape S, Vauloup-Fellous C, Morand-Joubert L, Roque-Afonso AM, Le Goff J, Delaugerre C. Evaluation of a Rapid Diagnostic Assay for Detection of SARS-CoV-2 Antigen in Nasopharyngeal Swabs. J Clin Microbiol. 2020 Jul 23;58(8):e00977-20. doi: 10.1128/JCM.00977-20. Print 2020 Jul 23. No abstract available. PMID 32404480
- [Background] Nagura-Ikeda M, Imai K, Tabata S, Miyoshi K, Murahara N, Mizuno T, Horiuchi M, Kato K, Imoto Y, Iwata M, Mimura S, Ito T, Tamura K, Kato Y. Clinical Evaluation of Self-Collected Saliva by Quantitative Reverse Transcription-PCR (RT-qPCR), Direct RT-qPCR, Reverse Transcription-Loop-Mediated Isothermal Amplification, and a Rapid Antigen Test To Diagnose COVID-19. J Clin Microbiol. 2020 Aug 24;58(9):e01438-20. doi: 10.1128/JCM.01438-20. Print 2020 Aug 24. PMID 32636214
- [Background] Castro R, Luz PM, Wakimoto MD, Veloso VG, Grinsztejn B, Perazzo H. COVID-19: a meta-analysis of diagnostic test accuracy of commercial assays registered in Brazil. Braz J Infect Dis. 2020 Mar-Apr;24(2):180-187. doi: 10.1016/j.bjid.2020.04.003. Epub 2020 Apr 18. PMID 32330437
- [Background] Mertens P, De Vos N, Martiny D, Jassoy C, Mirazimi A, Cuypers L, Van den Wijngaert S, Monteil V, Melin P, Stoffels K, Yin N, Mileto D, Delaunoy S, Magein H, Lagrou K, Bouzet J, Serrano G, Wautier M, Leclipteux T, Van Ranst M, Vandenberg O; LHUB-ULB SARS-CoV-2 Working Diagnostic Group. Development and Potential Usefulness of the COVID-19 Ag Respi-Strip Diagnostic Assay in a Pandemic Context. Front Med (Lausanne). 2020 May 8;7:225. doi: 10.3389/fmed.2020.00225. eCollection 2020. PMID 32574326
- [Background] Takeuchi Y, Akashi Y, Kato D, Kuwahara M, Muramatsu S, Ueda A, Notake S, Nakamura K, Ishikawa H, Suzuki H. Diagnostic performance and characteristics of anterior nasal collection for the SARS-CoV-2 antigen test: a prospective study. Sci Rep. 2021 May 18;11(1):10519. doi: 10.1038/s41598-021-90026-8. PMID 34006975
- [Background] Porte L, Legarraga P, Vollrath V, Aguilera X, Munita JM, Araos R, Pizarro G, Vial P, Iruretagoyena M, Dittrich S, Weitzel T. Evaluation of a novel antigen-based rapid detection test for the diagnosis of SARS-CoV-2 in respiratory samples. Int J Infect Dis. 2020 Oct;99:328-333. doi: 10.1016/j.ijid.2020.05.098. Epub 2020 Jun 1. PMID 32497809
- [Background] Mak GC, Cheng PK, Lau SS, Wong KK, Lau CS, Lam ET, Chan RC, Tsang DN. Evaluation of rapid antigen test for detection of SARS-CoV-2 virus. J Clin Virol. 2020 Aug;129:104500. doi: 10.1016/j.jcv.2020.104500. Epub 2020 Jun 8. PMID 32585619
- [Background] Blairon L, Wilmet A, Beukinga I, Tre-Hardy M. Implementation of rapid SARS-CoV-2 antigenic testing in a laboratory without access to molecular methods: Experiences of a general hospital. J Clin Virol. 2020 Aug;129:104472. doi: 10.1016/j.jcv.2020.104472. Epub 2020 May 30. PMID 32504944
- [Background] Scohy A, Anantharajah A, Bodeus M, Kabamba-Mukadi B, Verroken A, Rodriguez-Villalobos H. Low performance of rapid antigen detection test as frontline testing for COVID-19 diagnosis. J Clin Virol. 2020 Aug;129:104455. doi: 10.1016/j.jcv.2020.104455. Epub 2020 May 21. PMID 32485618
- [Background] Soleimani R, Deckers C, Huang TD, Bogaerts P, Evrard S, Wallemme I, Habib B, Rouze P, Denis O. Rapid COVID-19 antigenic tests: Usefulness of a modified method for diagnosis. J Med Virol. 2021 Sep;93(9):5655-5659. doi: 10.1002/jmv.27094. Epub 2021 May 31. PMID 34009649
- [Background] La Marca A, Capuzzo M, Paglia T, Roli L, Trenti T, Nelson SM. Testing for SARS-CoV-2 (COVID-19): a systematic review and clinical guide to molecular and serological in-vitro diagnostic assays. Reprod Biomed Online. 2020 Sep;41(3):483-499. doi: 10.1016/j.rbmo.2020.06.001. Epub 2020 Jun 14. PMID 32651106
- See also: Diagnosis of Acute Respiratory Syndrome Coronavirus 2 Infection by Detection of Nucleocapsid Protein — http://medrxiv.org/content/early/2020/03/13/2020.03.07.20032524.abstract

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Population: All subjects were aged 18 years or older and had symptoms consistent with COVID-19 (as assessed by their clinicians) for five days or less. All subjects underwent bilateral mid-turbinate swabs for COVID Antigen (Quidel Sofia SARS Antigen Fluorescent Immunoassay (FIA)) as well as bilateral rt-PCR testing (Quest SARS-CoV-2 rRT-PCR) via nasopharyngeal swab.
Period: Overall Study
Arm/Group | Study Population
Started | 117
Completed | 117
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Population
Number analyzed (Participants) | 117
Age, Customized [Count of Participants; unit: Participants] — Population: Age data were not collected for this study
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Gender data was not collected for this study
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 117

OUTCOME MEASURES:

1. Primary Outcome: Proportion of True Positives
Description: Of all Disease (rtPCR) Positive subjects, the proportion who were Test (antigen) Positive (sensitivity).
Time Frame: 1 day
Measure: Number (95% Confidence Interval); unit: proportion of true positives
Arm/Group | Study Population
Number analyzed (Participants) | 117
proportion of true positives | 0.750 [0.566 to 0.885]

2. Primary Outcome: Proportion of True Negatives
Description: Of all Disease (rtPCR) Negative subjects, the proportion who were Test (antigen) Negative (specificity).
Time Frame: 1 day
Measure: Number (95% Confidence Interval); unit: proportion of true negatives
Groups:
- Study Population: All subjects were aged 18 years or older and had symptoms consistent with COVID-19 (as assessed by their clinicians) for five days or less. No other baseline characteristics were collected.
Arm/Group | Study Population
Number analyzed (Participants) | 117
proportion of true negatives | 0.988 [0.936 to 1.000]

ADVERSE EVENTS:
Time Frame: 1 day
Description: The testing center staff/research coordinators were instructed to contact the Principal Investigator (or the Testing Center manager) for any unanticipated adverse events during the study. The details of the event would have been logged in RedCap. The risk of those events were to be assessed by the PI, appropriate medical care of the subject would have been ensured, and the IRB would have been informed of any event deemed more than minor, or for any event that recurred.
Arm/Group | Study Population
All-Cause Mortality (participants affected / at risk) | 0/117
Serious Adverse Events (participants affected / at risk) | 0/117
Other Adverse Events (participants affected / at risk) | 0/117

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT04610489/Prot_SAP_001.pdf